CLINICAL TRIAL: NCT01324856
Title: Results of Pancreaticogastrostomy Versus Pancreaticojejunostomy in Reconstruction After Cephalic Duodenopancreatectomy in Patients With Soft Pancreas and Small Pancreatic Duct
Brief Title: Pancreaticogastrostomy Versus Pancreaticojejunostomy in Reconstruction After Cephalic Duodenopancreatectomy
Acronym: PanAm
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Belgrade (Other)
Responsible Party: Dejan Radenkovic, Clinic for Digestive surgery, Clinical Center of Serbia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: D672
Record Dates: First submitted 2011-03-28; First posted 2011-03-29 (Estimated); Last update posted 2011-04-11 (Estimated); Status verified 2011-02

CONDITIONS: Pancreatic Cancer; Pancreatic Anastomotic Leak
Keywords: pancreatic cancer; periampulary cancer; pancreaticogastro vs pancreaticojejuno anastomosis
MeSH Terms: conditions — Pancreatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Pancreaticogastro anastomosis (Experimental)
  Interventions: Procedure: Pancreatico gastro anastomosis
- Pancreaticojejuno anastomosis (Active Comparator)
  Interventions: Procedure: Pancreaticojejuno anastomosis

INTERVENTIONS:
Procedure: Pancreatico gastro anastomosis — After the pylorus preserving cephalic pancreaticoduodenectomy, pancreatico gasto teremino-lateral anastomosis will be performed. The anastomosis will be done with posterior wall of the stomach. Pancreas will be mobilized at least 5 cm, two tobaco stiches will be applied on posterior wall of the stomach and hole of 2 cm will be done in the middle. Anterior wall of the stomach will be opened, for easier placement of the pancreas in to the stomach cavity. Pancreas will be entered in the stomach trough , tobacco stitches tided and just 2 or 3 stitches will be applied on the stomach mucosa and pancreatic capsule. After that classic hepatico jejuno and antecolic duodeno jejuno anatomosis will ber performed.
  Arms: Pancreaticogastro anastomosis
Procedure: Pancreaticojejuno anastomosis — After the pylorus preserving cephalic pancreaticoduodenectomy, pancreatico jejuno termino lateral duct to mucosa anastomosis will be performed. After that classic hepatico jejuno and antecolic duodeno jejuno anatomosis will ber performed.
  Arms: Pancreaticojejuno anastomosis

SUMMARY:
Pancreaticoduodenectomy is the standards surgical procedure for various malignant and benign disease of the pancreas and periampullariy region. During the recent years, mortality rate of pancreaticoduodenectomy has decreased to 5% in specialized centers. Although, this procedure still carries considerable morbidity up to 40%, depending of definition of complications. Pancreatic fistula remains a common complication and the main cause of other morbidities and mortality. Pancreaticojejunal (PJ) anastomosis is the most often used method of reconstruction after pancreaticoduodenectomy. Several technique modifications such as placement of the stents, reinforcement of anasomosis with fibrin glue, pancreatic duct occlusion and pancreaticogastrostomy (PG) type of anastomosis was used in order to decrease pancreatic fistula rate. Since, some retrospective studies showed better results with some technique, several meta-analyses did not show any advantage of those various modifications. It was shown that the higher risk of pancreatic fistula was noticed in patients with soft residual pancreas and small diameter of pancreatic duct. There is only one randomized study in the literature dealing with this problem. This study did not reveal any significant differences between PG and PJ in patients with soft pancreas and small duct. In order to investigate once more this important issue, the researchers conducted randomized multicenter controlled trial.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergone cephalic duodenopanceatectomy
* soft pancreas
* small diameter of the pancreatic remnant

Exclusion Criteria:

* Age bellow 18 and under 80
* prevous pancreatic surgery
* pregnancy
* Psychosis

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2011-04; Primary Completion 2013-04 (Estimated); Study Completion 2013-09 (Estimated)

PRIMARY OUTCOMES:
abdominal complications | 2 years
  Abdominal complications comprises: Pancreatic fistula, acute fluid collection, acute pancreatitis, billiay fistula, gastric fistula, enteral distula, hemorrhage and delayed gastric emptying

CONTACTS AND LOCATIONS:
Overall Officials: Dejan Radenkovic, MD,PhD, Principal Investigator — Clinic for Digestive disease, Clinical center of Serbia and School of Medicine University of Belgrade
Locations (4):
- Serbia (4):
  - Clinic for Digestive Surgery, Clinical Center of Serbia and School of Medicine University of Belgrade, Belgrade
  - Clinic for Emergency Surgery, Clinical Center of Serbia and School of Medicine, University of Belgrade, Belgrade
  - Surgical Department, Clinical Center "Bezanijska Kosa" and School of Medicine, University of Belgrade, Belgrade
  - Surgical Department, Military-Medical Academy, Belgrade

REFERENCES:
- [Background] Wente MN, Shrikhande SV, Muller MW, Diener MK, Seiler CM, Friess H, Buchler MW. Pancreaticojejunostomy versus pancreaticogastrostomy: systematic review and meta-analysis. Am J Surg. 2007 Feb;193(2):171-83. doi: 10.1016/j.amjsurg.2006.10.010. PMID 17236843
- [Background] Bassi C, Falconi M, Molinari E, Salvia R, Butturini G, Sartori N, Mantovani W, Pederzoli P. Reconstruction by pancreaticojejunostomy versus pancreaticogastrostomy following pancreatectomy: results of a comparative study. Ann Surg. 2005 Dec;242(6):767-71, discussion 771-3. doi: 10.1097/01.sla.0000189124.47589.6d. PMID 16327486
- [Background] Yeo CJ, Cameron JL, Maher MM, Sauter PK, Zahurak ML, Talamini MA, Lillemoe KD, Pitt HA. A prospective randomized trial of pancreaticogastrostomy versus pancreaticojejunostomy after pancreaticoduodenectomy. Ann Surg. 1995 Oct;222(4):580-8; discussion 588-92. doi: 10.1097/00000658-199510000-00014. PMID 7574936